CLINICAL TRIAL: NCT04395274
Title: Young Adult EC Use and Respiratory Outcomes
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alayna Tackett, Assistant Professor, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-23006; 1K01HL148907-01 (NIH); NCI-2024-06207 (Other: NCI)
Record Dates: First submitted 2020-04-21; First posted 2020-05-20 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: E Cig Use
Keywords: e-cigarette; respiratory health; prospective
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — salivary collection, respiratory health
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Current E-Cigarette Users: Monitoring current e-cigarette users
- Never E-Cigarette / Tobacco Users: Monitoring never users of any tobacco or e-cigarette products.

SUMMARY:
E-cigarette (EC) use continues to increase among youth, and EC may be detrimental to youth respiratory health. Public health officials and the Food and Drug Administration (FDA) can now regulate ECs. The proposed study uses naturalistic assessments called ecological momentary assessment (EMA) to understand how ECs use may impact the respiratory health of youth and young adult users compared to never-using peers.

DETAILED DESCRIPTION:
Using a prospective longitudinal design, 150 youth and young adults aged 18-25 years (100 exclusive-EC users; 50 never-users) will complete 5 sessions (baseline, 3-,6-, 9-, and 12-months). Sessions will include naturalistic measures such as measures of respiratory health, questionnaires, and nasal epithelial lining fluid (NELF) nasal samples. To assess acute changes in pulmonary functioning related to tobacco product use, participants will complete twice daily EMA and home-based spirometry for the 2 weeks following the Day 1 session and the 2 weeks prior to each follow-up zoom session. Never-users will participate in a brief 15-30-minute individual interview consisting of questions related to reasons for never-EC use and other protective factors that will be used to build future prevention messaging.

ELIGIBILITY:
Inclusion Criteria:

1. own a smartphone and willing to add study EMA and spirometry application to it.
2. a current exclusive-EC user (endorse ≥weekly use over the past 3 months) and report never trying OTPs
3. between the ages of 18-25 years old at the time of enrollment
4. read and speak English
5. willing to complete five, 2-week periods of daily EMA and home-based spirometry
6. never-users must indicate never trying any tobacco product to be eligible for enrollment

Exclusion Criteria:

1. self-reported diagnosis of lung disease including cystic fibrosis or chronic obstructive pulmonary disease; we will not exclude youth who have asthma, but will incorporate this as a covariate during analyses
2. unstable or significant psychiatric conditions (past and stable conditions will be allowed)
3. history of cardiac event or distress within the past 3 months
4. are currently pregnant, planning to become pregnant, or breastfeeding
5. are blind, severely visually impaired, deaf, hard of hearing, or have a severe motor disability

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The present proposal, a study of e-cigarette use among youth and young adults, will include both females and racial/ethnic minorities.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alayna Tackett, PhD, Principal Investigator — The Ohio State Comprehensive Cancer Center
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants are assigned to a study arm (Current E-Cigarette User or Never E-Cigarette/Tobacco User) after completion of the baseline survey. 10 Participants were found to be ineligible due to their tobacco use patterns reported at baseline, these participants were excluded from the study prior to being assigned to a study arm and are not included in the participant flow.
Period: Overall Study
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Started | 52 | 53
3-month | 26 | 46
6-month | 19 | 36
9-month | 12 | 34
12-month | 19 | 31
Completed | 19 | 31
Not Completed | 33 | 22
Not completed — Lost to Follow-up | 20 | 11
Not completed — Withdrawal by Subject | 13 | 10
Not completed — Moved Abroad | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only the 105 participants who were eligible at baseline are included. 10 participants were found to be ineligible after completing the baseline questionnaire.
Groups:
- Total: Total of all reporting groups
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.81 (2.11) | 20.11 (2.01) | 20.95 (2.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 45 | 74
  Male | 23 | 8 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 14 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 20 | 22 | 42
  More than one race | 6 | 7 | 13
  Unknown or Not Reported | 6 | 3 | 9
Days used e-cigarettes in past 30 days [Mean (Standard Deviation); unit: days] | 26.38 (6.24) | 0 (0) | 13.07 (13.96)

OUTCOME MEASURES:

1. Primary Outcome: Spirometry to Measure the Change From Baseline in Forced Vital Capacity (FVC)
Description: Participants will complete twice daily home-based spirometry (a pulmonary function diagnostic test) for the 2 weeks prior to each follow-up session.
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: Only participants who were eligible at baseline and provided spirometry measurements are included.
  The number of participants at follow-up is less than that at baseline due to loss to follow-up over time.
Measure: Mean (Standard Deviation); unit: liter
Units Other Than Participants: Forced Expiratory Maneuvers
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 43 | 49
Number analyzed (Forced Expiratory Maneuvers) | 780 | 1235
liter
  Baseline | 4.42 (1.30) | 3.54 (0.97)
  3-month: number analyzed (Participants) | 24 | 35
  3-month: number analyzed (Forced Expiratory Maneuvers) | 257 | 816
  3-month | 4.61 (1.70) | 3.68 (1.00)
  6-month: number analyzed (Participants) | 15 | 29
  6-month: number analyzed (Forced Expiratory Maneuvers) | 182 | 709
  6-month | 4.62 (1.66) | 3.96 (1.10)
  9-month: number analyzed (Participants) | 8 | 25
  9-month: number analyzed (Forced Expiratory Maneuvers) | 161 | 597
  9-month | 4.52 (1.26) | 3.89 (1.09)
  12-month: number analyzed (Participants) | 18 | 30
  12-month: number analyzed (Forced Expiratory Maneuvers) | 295 | 738
  12-month | 4.34 (1.45) | 4.33 (1.00)

2. Primary Outcome: Spirometry to Measure the Change From Baseline in Forced Expiratory Volume (FEV)
Description: as for outcome 1
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Units Other Than Participants: Forced Expiratory Maneuvers
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 43 | 49
Number analyzed (Forced Expiratory Maneuvers) | 780 | 1235
Liters
  Baseline | 3.63 (0.93) | 3.04 (0.70)
  3-month: number analyzed (Participants) | 24 | 35
  3-month: number analyzed (Forced Expiratory Maneuvers) | 257 | 816
  3-month | 3.64 (1.12) | 3.18 (0.72)
  6-month: number analyzed (Participants) | 15 | 29
  6-month: number analyzed (Forced Expiratory Maneuvers) | 182 | 709
  6-month | 3.67 (1.15) | 3.36 (0.83)
  9-month: number analyzed (Participants) | 8 | 25
  9-month: number analyzed (Forced Expiratory Maneuvers) | 161 | 597
  9-month | 3.81 (0.85) | 3.34 (0.84)
  12-month: number analyzed (Participants) | 18 | 29
  12-month: number analyzed (Forced Expiratory Maneuvers) | 295 | 738
  12-month | 3.60 (0.96) | 3.63 (0.82)

3. Primary Outcome: Level of Dependence by Product Type Will be Examined.
Description: Changes in product use evaluated with an evaluation of the changes in dependence using the Hooked on Nicotine Checklist (HONC).
  Scores range from 0 to 10 with higher values indicating greater levels of dependence.
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: Only participants who were eligible and using e-cigarettes at baseline are included.
  The number of participants at follow-up is less than that at baseline due to loss to follow-up over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Disposable Users: Current e-cigarette users who report a disposable vape as being their main vaping device
- Pod Mod Users: Current e-cigarette users who report a pod mod as being their main vaping device
- Other Device Type Users: Current e-cigarette users who report a device other than a disposable or pod mod as being their main vaping device
Arm/Group | Disposable Users | Pod Mod Users | Other Device Type Users
Number analyzed (Participants) | 24 | 20 | 6
score on a scale
  Baseline | 5.83 (3.06) | 7.35 (2.83) | 7.67 (2.34)
  3-month: number analyzed (Participants) | 11 | 9 | 2
  3-month | 5.55 (3.36) | 8.44 (1.01) | 7.00 (1.41)
  6-month: number analyzed (Participants) | 10 | 6 | 0
  6-month | 6.30 (3.71) | 8.50 (1.38) |
  9-month: number analyzed (Participants) | 7 | 3 | 0
  9-month | 5.86 (3.08) | 8.33 (0.58) |
  12-month: number analyzed (Participants) | 7 | 5 | 0
  12-month | 6.71 (3.35) | 7.40 (0.89) |

4. Primary Outcome: Respiratory Health Measures by Nasal Swab - IL-6
Description: Nasal epithelial lining fluid (NELF) samples will provide objective data on respiratory health (e.g., markers of inflammation, host defense, and lung injury) and will provide estimates of nicotine exposure/use via cotinine (i.e., the predominate metabolite of nicotine).
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: The population of participants who both attended their study visit and were able to provide a NELF sample is analyzed. Note that not all participants provided a sample at all visits.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 14.31 (24.97) | 9.95 (19.57)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 49.50 (113.35) | 17.63 (35.50)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 19.72 (30.59) | 37.01 (91.92)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 14.83 (27.87) | 12.63 (25.82)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 11.16 (19.36) | 48.85 (141.49)

5. Primary Outcome: Respiratory Health Measures by Nasal Swab - IL-8
Description: Nasal epithelial lining fluid (NELF) samples will provide objective data on respiratory health (e.g., markers of inflammation, host defense, and lung injury) and will provide estimates of nicotine exposure/use via cotinine (i.e., the predominate metabolite of nicotine) will also be examined to provide objective indicators of recency of EC and/or OTP use.
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 6637.06 (10518.30) | 12872.08 (23804.68)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 7630.32 (13048.51) | 13890.15 (21078.75)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 9509.56 (18926.62) | 20161.25 (57400.44)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 13648.62 (17464.65) | 16718.97 (20585.58)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 5071.09 (5763.48) | 13701.80 (22627.42)

6. Primary Outcome: Respiratory Health Measures by Nasal Swab - TNF-alpha
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 5.86 (6.87) | 4.98 (5.07)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 11.14 (14.83) | 7.15 (8.12)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 6.53 (5.32) | 6.25 (6.31)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 8.15 (7.31) | 6.53 (7.35)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 6.31 (6.81) | 11.52 (26.98)

7. Primary Outcome: Respiratory Health Measures by Nasal Swab - IL-4
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 0.46 (1.48) | 0.12 (0.17)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 0.34 (0.41) | 0.38 (1.08)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 0.12 (0.16) | 0.23 (0.26)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 0.19 (0.23) | 0.21 (0.25)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 0.13 (0.16) | 0.32 (0.49)

8. Primary Outcome: Respiratory Health Measures by Nasal Swab - IL-5
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 7.45 (24.78) | 0.64 (1.61)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 8.10 (24.75) | 0.58 (1.43)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 2.40 (5.13) | 1.79 (7.11)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 1.12 (1.51) | 0.48 (0.97)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 1.29 (1.87) | 6.16 (15.55)

9. Primary Outcome: Respiratory Health Measures by Nasal Swab - IL-10
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 3.17 (14.95) | 0.75 (0.86)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 16.73 (70.79) | 1.41 (2.11)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 2.10 (4.12) | 46.13 (250.36)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 0.91 (1.14) | 0.90 (1.25)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 55.95 (238.43) | 47.67 (255.71)

10. Primary Outcome: Respiratory Health Measures by Nasal Swab - IL-13
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 14.68 (14.63) | 13.13 (9.31)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 16.94 (11.52) | 16.02 (14.30)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 14.02 (9.01) | 14.28 (10.80)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 20.17 (13.70) | 15.49 (13.59)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 13.70 (11.85) | 19.25 (18.24)

11. Primary Outcome: Respiratory Health Measures by Nasal Swab - TARC
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 8.97 (11.59) | 26.73 (38.79)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 16.88 (24.04) | 41.36 (83.93)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 19.28 (34.76) | 26.22 (24.10)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 17.37 (22.86) | 26.11 (22.82)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 27.19 (63.00) | 68.70 (195.73)

12. Primary Outcome: Respiratory Health Measures by Nasal Swab - Eotaxin
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 135.72 (145.29) | 167.33 (214.22)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 135.21 (122.14) | 208.15 (223.99)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 228.79 (236.56) | 188.60 (252.67)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 191.06 (120.87) | 206.17 (258.11)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 234.12 (290.53) | 220.85 (226.80)

13. Primary Outcome: Respiratory Health Measures by Nasal Swab - MCP-1
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 198.65 (186.20) | 228.50 (205.86)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 247.34 (407.93) | 387.24 (454.32)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 316.92 (274.02) | 289.26 (254.87)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 284.78 (139.83) | 371.59 (446.76)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 255.77 (193.15) | 299.07 (308.34)

14. Primary Outcome: Respiratory Health Measures by Nasal Swab - MCP-4
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 49
pg/mL
  Baseline | 6.88 (10.71) | 6.94 (11.50)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 5.94 (7.21) | 7.79 (10.28)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 16.62 (32.59) | 8.74 (19.83)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 9.79 (9.46) | 6.27 (10.51)
  12-month: number analyzed (Participants) | 19 | 31
  12-month | 8.93 (12.11) | 8.07 (9.99)

15. Primary Outcome: Respiratory Health Measures by Nasal Swab - Cotinine
Description: as for outcome 5
Time Frame: Baseline, 3-month, 6-month, 9-month, 12-month
Population: The population of participants who both attended their study visit and were able to provide a sample is analyzed. Note that not all participants provided a sample at all visits.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
Number analyzed (Participants) | 42 | 50
ng/mL
  Baseline | 156.56 (162.53) | 0.09 (0.13)
  3-month: number analyzed (Participants) | 23 | 38
  3-month | 145.43 (129.93) | 0.08 (0.00)
  6-month: number analyzed (Participants) | 15 | 32
  6-month | 146.15 (165.97) | 0.09 (0.08)
  9-month: number analyzed (Participants) | 9 | 25
  9-month | 195.47 (190.39) | 0.07 (0.00)
  12-month: number analyzed (Participants) | 18 | 31
  12-month | 163.56 (233.97) | 6.83 (37.63)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Current E-Cigarette Users | Never E-Cigarette / Tobacco Users
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 11/52 | 0/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Current E-Cigarette Users (N=52) | Never E-Cigarette / Tobacco Users (N=53)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Sore or dry mouth and throat (General disorders) | 5 | 0
Headache (General disorders) | 4 | 0
Dizziness (General disorders) | 2 | 0
Sleepiness (General disorders) | 3 | 0
Sleeplessness (General disorders) | 2 (3) | 0
Heart palpitations (Cardiac disorders) | 1 | 0
Breathing difficulties (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Shortness of breath (General disorders) | 6 | 0
Allergies (Immune system disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Nausea (General disorders) | 2 | 0
Throat tightness (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT04395274/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT04395274/SAP_001.pdf